CLINICAL TRIAL: NCT01934465
Title: Assessment of Clinical Practice Administration of Chemotherapy and Anti-angiogenic Agent (Bevacizumab) Retrospectively and Prospectively as First Line Treatment for Patients With Advanced or Metastatic Non Small Cell Lung Cancer. Assessment of Toxicity, Compliance and Survival of Patients.
Brief Title: Bevacizumab Plus Chemotherapy for Advanced Non Small Cell Lung Cancer Patients as 1st Line Treatment
Status: Completed | Type: Observational
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CT/10.11
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Chemotherapy; Anti-angiogenic agent; Bevacizumab; 1st Line
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Avastin regimens: Patients who have either received or who are going to receive chemotherapy plus Avastin (bevacizumab)

SUMMARY:
Investigators propose to assess, retrospectively and prospectively the safety and tolerability profile (number of participants with adverse events) of standard chemotherapy and anti-angiogenic agent bevacizumab (Avastin) as first line treatment of patients with advanced or metastatic Non Small Cell Lung Cancer.

All treatment schedules that are going to be assessed are considered by the international guidelines as standard therapy for patients with advanced or metastatic Non Small Cell Lung Cancer.

DETAILED DESCRIPTION:
In addition investigators propose to assess the compliance of patients to treatment and the efficacy of treatment. That means percentage of objective responses, duration of response, progression free survival and estimation of overall survival

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any trial-specific procedure or treatment
* Ability to comply with the protocol
* Histologically or cytologically (sample to be obtained by biopsy or bronchoscopy) confirmed non-squamous NSCLC (locally recurrent or metastatic) per investigator assessment
* At least 1 unidimensionally measurable lesion meeting RECIST criteria
* No prior first line treatment for metastatic colorectal cancer
* Age ≥18 years
* ECOG performance status ≤2
* Adequate haematological, renal and hepatic function
* Urine protein <2+ (dipstick)
* International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN within 7 days prior to randomization, unless there is prophylactic use of anti-coagulation
* Patients with asymptomatic treated brain metastases are eligible for trial participation. Patients must complete treatment for brain metastases (radiotherapy with or without surgery, or stereotactic radiosurgery), including steroids, at least 28 days prior to randomization. Treatment with anticonvulsants at the time of randomization (i.e. ≥ 28 days) is allowed as long as the anti-convulsant is at a stable dose)
* Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as >2 years after last menstruation or surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, i.e. with a failure rate of less than 1% per year, are implants, injectables, combined oral contraceptives, intra-uterine device [IUD; only hormonspirals], sexual abstinence or vasectomized partner) during the trial and for a period of at least 6 months following the last administration of trial drug(s).Female patients with an intact uterus (unless amenorrhoeic for the last 24 months) must have a negative serum pregnancy test within 7 days prior to randomization into the trial
* Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control, i.e. with a failure rate of less than 1% per year, include a female partner using implants, injectables, combined oral contraceptives, IUDs [only hormonspirals], sexual abstinence or prior vasectomy) during the trial and for a period of at least 6 months following the last administration of trial drug(s)

Exclusion Criteria:

* Mixed, non-small cell and small cell tumors or mixed adenosquamous carcinomas with a predominant squamous component
* History of hemoptysis ≥ grade 2 (defined as bright red blood of at least 2.5 mL) within 3 months prior to randomization
* Surgery (including open biopsy), significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during trial treatment
* Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion
* Evidence of tumor invading or abutting a major blood vessel (e.g., pulmonary artery or superior vena cava) on imaging
* Radiotherapy to any site for any reason within 28 days prior to randomization. Palliative radiotherapy to bone lesions within 14 days prior to randomization is allowed
* Current or recent (within 10 days prior to first dose of bevacizumab) use of aspirin (> 325 mg/day), clopidogrel (> 75 mg/day), or current or recent (within 10 days prior to first dose of bevacizumab) use of full-dose (i.e. therapeutic dose) oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes. Prophylactic use of anticoagulants is allowed.
* History or evidence of inherited bleeding diathesis or coagulopathy with a risk of bleeding
* Active gastrointestinal bleeding
* Inadequately controlled hypertension (blood pressure: systolic > 150 mmHg and/or diastolic > 100 mmHg) within 28 days prior to randomization or history of hypertensive crisis or hypertensive encephalopathy
* Clinically significant (i.e. active) cardiovascular disease (e.g. cerebrovascular accident [CVA] or myocardial infarction within 6 months prior to randomization, unstable angina, congestive heart failure [CHF] New York Heart Association [NYHA] Class ≥ II, or serious cardiac arrhythmia), that is uncontrolled by medication or may interfere with administration of trial treatment
* Non-healing wound, active peptic ulcer or untreated bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra abdominal abscess within 6 months prior to randomization.
* Treatment with any other investigational agent within 28 days prior to randomization. Patients in the follow-up phase of 1st-line trials who fulfill all eligibility criteria may be enrolled in this trial if the 1st-line protocol allows bevacizumab-based treatment in the follow-up phase
* Known hypersensitivity to bevacizumab or any of its excipients, or any of the SOC agents foreseen
* Malignancy other than NSCLC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent, and ductal carcinoma in situ (DCIS) treated surgically with curative intent
* Evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational or SOC drug used in this study or puts the patient at higher risk for treatment-related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics for cancer prevention
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with AE | Every 3 weeks up to 18 weeks
  In this observational study investigators are going to assess standard schedules in which administrations were every 3 weeks.

SECONDARY OUTCOMES:
Number of Participants with Response Rate | Disease evaluation at Week 6
  In this observational study investigators are going to assess standard schedules in which the disease evaluation was performed every 6 weeks
Percentage of Patients with Progression Free Survival | 1 year
Patients Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — Hellenic Oncology Research Group
Locations (8):
- Greece (8):
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dept. of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Matikas A, Kentepozidis Nu, Ardavanis A, Vaslamatzis M, Polyzos A, Emmanouilides Ch, Katsaounis P, Koinis F, Xynogalos S, Christopoulou A, Ziras N, Tegos T, Prinarakis E, Hatzidaki D, Georgoulias V, Kotsakis A; HORG's Lung Cancer Working Group. Efficacy and tolerance of frontline bevacizumab-based chemotherapy for advanced non-small cell lung cancer patients: a multicenter, phase IV study of the Hellenic Oncology Research Group (HORG). Cancer Chemother Pharmacol. 2016 Aug;78(2):369-76. doi: 10.1007/s00280-016-3094-7. Epub 2016 Jun 22. PMID 27335027